CLINICAL TRIAL: NCT03366350
Title: A Phase 1/2 Study Evaluating the Safety and Efficacy of Anti-CD19 Chimeric Antigen Receptor-Modified T Cell (CAR-T) Therapy Bridging to Hematological Stem Cell Transplantation (HSCT) for Relapsed/Refractory CD19+ B-Cell Malignancies
Brief Title: Anti-CD19 CAR-T Therapy Bridging to HSCT for CD19+ B-Cell Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuhan Sian Medical Technology Co., Ltd (Industry)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Jingzhou Central Hospital (Other); Xiangyang Central Hospital (Other); People Hospital Of Yichang (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CART-CD19-02
Record Dates: First submitted 2017-12-01; First posted 2017-12-08 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Acute Lymphoblastic Leukemia; B Cell Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, B-Cell

STUDY DESIGN:
Intervention Model Description: Patients receive consolidative allo-HSCT following CAR-T therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Consolidative allo-HSCT following CAR-T therapy (Experimental): Patients who had achieved MRD-negative complete remissions through CAR-T therapy (NCT02965092) will, on their own accord, receive allo-HSCT if there are no previous HSCT, contraindications, and other restrictions.
  Interventions: Procedure: Allogeneic hematological stem cell transplantation

INTERVENTIONS:
Procedure: Allogeneic hematological stem cell transplantation — Patients receive allogeneic hematological stem cell transplantation after they achieve MRD- CR through CAR-T therapy.

SUMMARY:
This is the second stage of the previous anti-CD19 CAR-T therapy (NCT02965092). The study aims to evaluate the safety and efficacy of consolidative allo-HSCT following CAR-T therapy in patients with relapsed or refractory B cell Malignancies.

DETAILED DESCRIPTION:
Anti-CD19 CAR-T therapy has been confirmed effective for relapsed/refractory B-cell malignancies. However, its ability to keep patients in maintained remission is limited. In order to keep patients in long-term remissions, patients who had achieved MRD-negative complete remissions through CAR-T therapy (NCT02965092) will, on their own accord, receive allo-HSCT if there are no previous HSCT, contraindications, and other restrictions.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is pathologically and histologically confirmed as CD19 + B cell malignancies, and has achieved MRD-negative CR through CAR-T therapy (NCT02965092);
2. B cell hematological malignancies include the following three categories:

   * B-cell acute lymphocytic leukemia (B-ALL);
   * Indolent B-cell lymphoma (CLL, FL, MZL, LPL);
   * Aggressive B-cell lymphoma (DLBCL, BL, MCL);
3. < 70 years old;
4. Expected survival time > 6 months;
5. Female patients around childbearing age, negative pregnancy test before trial, and agreed to take effective contraceptive measures during the trial until the last visit;
6. Voluntarily participate in this experiment and sign informed consent by themselves, or legally authorized representative.

Exclusion Criteria:

1. With a history of epilepsy or other central nervous system diseases;
2. Previous allogeneic hematopoietic stem cell transplantation;
3. The presence of clinically significant cardiovascular disease, such as uncontrolled or symptomatic arrhythmias, congestive heart failure or myocardial infarction within recent six months, or heart disease with cardiac function in any grade 3 (moderate) or 4 ( severe) (according to the New York Heart Association (NYHA) Functional Classification System);
4. Pregnant or lactating women (safety of this therapy for the unborn child is unknown);
5. Not curable active infection;
6. Patients with active hepatitis B or hepatitis C virus infection;
7. Combined use of systemic steroids within two weeks (except use of inhaled steroid recently or currently);
8. Creatinine> 2.5 mg / dl (221.0 umol/L); ALT / AST> 3 X the normal amount; Bilirubin> 2.0 mg / dl (34.2 umol/L);
9. Patients suffering from other uncontrolled diseases, and researchers believe that the patient is not suitable for trial;
10. Patients with HIV-infection;
11. Any situation that may increase the risk of patients or interfere with test results.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-04-15 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 5 years
  To evaluate the safety of anti-CD19 CAR-T therapy bridging to allo-HSCT. Therapy-related adverse events were recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 4.0)

SECONDARY OUTCOMES:
Overall survival | 5 years
  OS was calculated from the date of inclusion to death or last follow-up (censored).
Event-free survival | 5 years
  EFS was calculated from the date of inclusion to death, progression of the disease, relapse or gene recurrence, whichever came first, or last visit (censored).
Relapse-free survival | 5 years
  RFS was calculated from the date of inclusion to relapse or last visit (censored).

CONTACTS AND LOCATIONS:
Overall Officials: YU HU, M.D., Ph.D, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Du M, Mayombo RTM, Liu J, Zhang Y, Liao D, Hu Y, Mei H. The impact of obesity and its related underlying diseases on cytokine release syndrome and the efficacy of CAR-T therapy in treating B-cell malignancies. Ann Hematol. 2025 Mar;104(3):1887-1895. doi: 10.1007/s00277-025-06338-6. Epub 2025 Apr 8. PMID 40195173